CLINICAL TRIAL: NCT06192641
Title: Benefits of Melatonin Use in Patients With Climacterious Symptoms in the Perimenopause: Randomized, Double-blind, Placebo-controlled Clinical Trial
Brief Title: Melatonin Use in Patients With Climacterious Symptoms in the Perimenopause
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Univates (Other)
Collaborators: Aline Patrícia Brietzke (Unknown); Ana Paula Costella (Unknown)
Responsible Party: Principal Investigator, Gabriela Laste, Professor, Univates
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10901364
Record Dates: First submitted 2023-12-19; First posted 2024-01-05 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Perimenopausal Disorder
MeSH Terms: interventions — Melatonin

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, parallel, placebo-controlled clinical trial. 40 patients will be recruited to participate in the study, 20 of whom will receive the treatment and 20 will receive the placebo.Patients will receive 3 mg melatonin in capsule or placebo (capsule identical to the treatment, both in color, taste, odor and shape, composed of cellulose and indigestible fiber) (PALMER, 2020). (GOLTZMAN, 2021) for 30 days (Treister-Goltzman; Peleg, 2021) They will be instructed to ingest melatonin once a day, at night, one hour before bed (PALMER, et al. 2020).
Who Masked: Participant, Investigator
Masking Description: To control possible measurement biases, in the present study, the following measures will be taken: for the pharmacological intervention (use of melatonin or placebo), the evaluators and patients will be blinded to the intervention. The randomization codes will remain in the care of two evaluators not involved in the care of the patients, which allows better control of manipulations to favor any intervention to be carried out. Patients will be instructed to discuss all aspects related to pharmacological interventions with the researcher during treatment. The sealed envelope method will be used for confidential allocation. Before the recruitment phase, envelopes containing protocol materials will be prepared. Each envelope containing the allocated treatment will be sealed and numbered sequentially. After each participant agrees to participate in the study, the envelope will be opened and the results will be reported to the researcher who will carry out the interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Melatonin (Active Comparator): Patients will receive 3 mg melatonin in capsule for 30 days. They will be instructed to ingest melatonin once a day, at night, one hour before bed.
  Interventions: Drug: Melatonin 3 MG
- Placebo (Placebo Comparator): Patients will receive placebo capsule composed of cellulose and indigestible fiber for 30 days. They will be instructed to ingest melatonin once a day, at night, one hour before bed.
  Interventions: Drug: Melatonin 3 MG

INTERVENTIONS:
Drug: Melatonin 3 MG — patients received 3 mg melatonin in capsule or placebo (capsule identical to the treatment, both in color, taste, odor and shape, composed of cellulose and indigestible fiber) (PALMER, 2020). (GOLTZMAN, 2021) for 30 days (Treister-Goltzman; Peleg, 2021) They will be instructed to ingest melatonin once a day, at night, one hour before bed (PALMER, et al. 2020).
  Other Names: melatonin

SUMMARY:
Menopause is defined as the absence of menstruation for 12 months without a pathological cause and it is marked by physical fluctuations and biological changes that can impact women's quality of life. During the perimenopause and menopause transition period, women may experience a variety of changes, including menstrual cycle irregularity and climacteric symptoms. Treatment to relieve symptoms may include hormonal and non-hormonal options, such as behavioral therapies, medications and low-dose hormonal therapies. The objective of this study will be to evaluate the effect of melatonin in women with perimenopausal symptoms. This is a double-blind, placebo-controlled randomized clinical trial research, where perimenopausal women will be interviewed, who will answer questionnaires, and will use melatonin/placebo for a period of 30 days, before and after, they will be asked about possible changes during treatment, such as mood changes, drowsiness, dizziness, headaches or allergic reactions. It is hoped that with this study, the effect of melatonin in women on climacteric symptoms during the perimenopausal period will be understood.

DETAILED DESCRIPTION:
This is a randomized, double-blind, parallel, placebo-controlled clinical trial. 40 patients will be recruited to participate in the study, 20 of whom will receive the treatment and 20 will receive the placebo for a period of 30 days.Before and after, they will be asked about possible changes during treatment, such as mood changes, drowsiness, dizziness, headaches or allergic reactions.

The study will be carried out at the São Cristóvão Basic Health Unit in Lajeado - RS. The research and invitation to participate will also be publicized through the University of Vale do Taquari's social media, through an informative/explanatory text. Data collection from these participants will be carried out at their homes or in a location that suits them best by arrangement. If the participant has travel expenses for their participation, travel/transportation costs will be reimbursed within the project budget, which will be the responsibility of the responsible researcher.

The study protocol was submitted and approved by the Univates Health Research Ethics Committee by CAAE: 70400923.9.0000.5310 and opinion no.: 6.131.475.

For statistical analyzes the statistical program JAMOVI (Version 2.3) [Computer Software] (2022) and R Core Team (2021) will be used. The Kolmogorov Smirnov and Shapiro-Wilk Test will be used to verify the normality of the data. Non-parametric samples will be analyzed using the Mann-Whitney U test and parametric t-test. Continuous variables will be presented as mean±SD. The number and percentage will be presented as n (%), and numerical data will be analyzed using the Chi-square test (χ²) and/or Fisher's exact test. The Confidence Interval value (IC95%) will be provided. The value of p<0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:- Being female and in peri-menopause, experiencing an irregular menstrual cycle, having had at least one menstrual period in the last 6 months.

* Age 45 years or older
* Be literate

Exclusion Criteria:-History of alcohol or other substance abuse in the last 6 months

* Use of hormonal therapy;
* Neurological disease;
* Oncological disease;
* Ischemic heart disease;
* Liver failure;
* Renal insufficiency;
* Use of central nervous system medications (antidepressants, anticonvulsants, antipsychotics and benzodiazepines)

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-10-20 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Menopause rating scale | one month
  Menopause scale, 0-44, higher score worse outcome

SECONDARY OUTCOMES:
Beck Depression Inventory II | one month
  Level of depressive symptoms, 0-63, higher score worse outcome. Score 16 is considered depression.
Pittsburgh Sleep Quality Index | one month
  Sleep quality, 0-20, higher score worse sleep
Visual Analog Pain Scale | daily for one month
  pain scale, can vary from zero (no pain) to 100 mm (worst possible pain)
Hamilton scale | one month
  anxiety rating scale, 0-56, >30 severe anxiety.
Visual analogue scale of sleep | daily for one month
  sleep scale, varies from worst possible (0) to best possible (10 cm)

CONTACTS AND LOCATIONS:
Locations (1):
- Gabriela Laste, Lajeado, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No